CLINICAL TRIAL: NCT04937348
Title: Visfatin and Omentin-1 - Markers of Nutritional Status of Newborns Born to Diabetic Mothers.
Status: Completed | Type: Observational
Sponsor: Wroclaw Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 773/2019; STM.A300.20.143 (Other Grant/Funding Number: Wroclaw Medical University)
Record Dates: First submitted 2021-06-11; First posted 2021-06-24 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2021-05

CONDITIONS: Gestational Diabetes; Diabetes Mellitus; Neonate; Nutritional Status
Keywords: gestational diabetes; adipokines; visfatin; omentin; nutritional status; neonate; breast milk
MeSH Terms: conditions — Diabetes, Gestational; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum, breast milk
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- GDM G1: Mothers diagnosed with gestational diabetes mellitus, treated with diet; and their newborns
  Interventions: Diagnostic Test: Acquisition and analysis of milk samples; Diagnostic Test: Collection, preparation and analysis of mother's blood samples.; Diagnostic Test: Body composition assessment; Other: Anthropometric measurements
- GDM G2: Mothers diagnosed with gestational diabetes mellitus, treated with insulin; and their newborns
  Interventions: Diagnostic Test: Acquisition and analysis of milk samples; Diagnostic Test: Collection, preparation and analysis of mother's blood samples.; Diagnostic Test: Body composition assessment; Other: Anthropometric measurements
- non-GDM / control group: Healthy, non-diabetic mothers, without disturbances in glucose metabolism; and their newborns.
  Control group.
  Interventions: Diagnostic Test: Acquisition and analysis of milk samples; Diagnostic Test: Collection, preparation and analysis of mother's blood samples.; Diagnostic Test: Body composition assessment; Other: Anthropometric measurements

INTERVENTIONS:
Diagnostic Test: Acquisition and analysis of milk samples — In order to ensure reproducible results, breast milk samples were collected using a breast pump. Samples were taken in the morning, after the newborn was breastfed. The entire breast was emptied. In order to ensure the stability of the microbiological and nutritional composition, the milk samples were cooled immediately after collection, and then divided into test tubes and frozen (-80 C) until the laboratory tests were made.
  The concentrations of macronutrients (protein, fat, carbohydrate) in breast milk were determined using a Human Milk Analyzer (HMA; Miris, Uppsala). Tissue hormones, e.g. adipokines: visfatin, omentin-1 were determined by ELISA method using commercial reagent kits.
Diagnostic Test: Collection, preparation and analysis of mother's blood samples. — Blood samples were collected from the mothers (fasting if possible) on the day the milk samples were taken. After collection, fasting glucose and insulin, as well as glycated hemoglobin were marked, and the other samples were centrifuged and frozen until analyzed (-80 C). Determination of adipokines was performed by ELISA method, using commercial reagent kits.
Diagnostic Test: Body composition assessment — The body composition of newborns was determined by a non-invasive electrical bioimpedance method using the body composition analyzer.
Other: Anthropometric measurements — Based on the mother's medical records, maternal height and pregnancy weight changes were recorded. On the day the biological material is collected, the mother was weighed.
  From the baby's documentation, measurements of the length, head circumference and body weight taken after delivery and during the hospitalization were recorded. These measurements were repeated on the days of the body composition analysis.

SUMMARY:
Diabetes mellitus is one of the most common metabolic disorders complicating the course of pregnancy, which concerns pre-pregnancy diabetes (PGDM) - most often type 1 or type 2; and gestational diabetes (GDM) - treated with diet (G1) or insulin (G2). Currently, in the pathogenesis of diabetes and the regulation of glucose metabolism, the role of tissue hormones, including adipokines, e.g., omentin-1, visfatin, have been considered. Adipokines might also affect the development of the fetus - mainly fetal adipose tissue gain. Their concentrations and activity depend on the maternal visceral fat content and concomitant metabolic disorders. It is known that adipokines are excreted in human milk during the lactation period.

The aim of the study was to assess the impact of diabetes during pregnancy, requiring treatment with diet or insulin, on the nutritional status of the newborn.

DETAILED DESCRIPTION:
The detailed aim of the study was to analyze the relationship between the concentration of selected adipokines, visfatin and omentin-1 in the mother, and the nutritional status of the newborn (expressed as body composition and anthropometric measurements), as well as the composition of breast milk, and clinical data on the course of pregnancy, childbirth, puerperium (interview from mother) and the postnatal stay of the child in the hospital.

Primary protocol:

The research was going to be conducted twice, that is:

1. in the period of postnatal hospitalization of the newborn, before discharge from the hospital (up to 7 days of age) in the Neonatology Clinic,
2. in the 4th - 6th week of the child's life, after visiting the Neonatology Outpatient Clinic.

Apart from the clinical examination, anthropometric measurements and body composition measurements, the results of laboratory tests performed on a child during hospitalization up to the 7th day of life and at the 4-6 week of life were collected. The interview questionnaire was carried out twice with the child's mother. From the mother, at the same time, milk (colostrum and mature) and blood was collected for laboratory tests.

Further changes in the protocol (accepted by Bioethical Comitte):

1. Extending the project with further study visits, i.e. 6-12 weeks and if the mother wishes to continue participation, 13 weeks - 6 months after delivery, in the case of sustained lactation and further breastfeeding, before introducing solid food into the child's diet.

   Substantiation: Due to the COVID-19 pandemic, the second project visit was abandoned. Based on telephone calls, the patients were still interested in participating, the more so as they had not completed the prescribed postpartum check-ups, their scheduled visits to specialists were canceled, and the infant vaccinations had been postponed. Patients also reported the need for lactation advice. Additional dates (6-12 weeks after childbirth and 13 weeks to 6 months after childbirth) would enable inviting mothers and their babies, providing medical or lactation advice according to their needs, as well as continuing the project among patients and their children who had been included in the study so far.
2. Cooperation with Biobank of Wrocław Medical University was established.

Substantiation: Possibility of collecting and storing biological material for further research in safe and controlled conditions.

ELIGIBILITY:
Inclusion Criteria:

* mother's age 18 - 45 years;
* delivery at term (≥ 37 + 0/7 weeks of pregnancy) or close to the delivery date (from 35 + 0/7 to 36 + 6/7 weeks of pregnancy), both by vaginal delivery and by caesarean section;
* single pregnancy;
* good condition of the child after birth, rated > 7 points on the Apgar score after the 1 st minute of life;
* feeding the baby only naturally (with breast or expressed breast milk) or mainly naturally;
* mother's informed and voluntary consent to participate in the study;
* mother's informed and voluntary consent to the participation of her child in the study.

Exclusion Criteria:

* mother's lack of consent to participate in the study;
* mother's lack of consent to the participation of her child in the study;
* mother's age <18 years and > 45 years;
* preterm labor <35 + 0/7 weeks of pregnancy;
* multiple pregnancy;
* the child's condition at birth is moderate or severe, rated at ≤ 7 points on the Apgar score after the 1st minute of life;
* feeding a child exclusively or mainly with an infant formula;
* severe birth defects of a newborn,
* any clinical condition of the mother and / or the newborn that may affect the nutritional status of the newborn (IUGR, lack of medical care during pregnancy, addiction of the mother to alcohol or other psychoactive substances, nicotinism in pregnancy, uncontrolled asthma in the mother, metabolic diseases in the mother or newborn).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study group included mothers with diagnosed diabetes and their newborns. Women with gestational diabetes, both treated with diet and treated with insulin - each group was supposed to include at least 20 patients. Additionally, if possible, women diagnosed with type 1 and type 2 pre-pregnancy diabetes or insulin resistance might have been included in the study. The control group consisted of 20 healthy women and their newborns.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2019-12-13 (Actual); Primary Completion 2021-02-05 (Actual); Study Completion 2021-03-17 (Actual)

PRIMARY OUTCOMES:
Fat body mass [kg] | up to 6 months
  Changes in infantile fat body mass between 2 timepoints (the first week of life and the 2nd visit).
Total body water [l] | up to 6 months
  Changes in infantile total body water between 2 timepoints (the first week of life and the 2nd visit).
Anthropometrics: body weight [kg], length [cm], head circumference [cm]. | up to 6 months
  Changes in infantile anthropometrics between 2 timepoints (the first week of life and the 2nd visit). On the basis of weight and length, BMI (kg/m2) and Ponderal Index will be calculated (kg/m3).

SECONDARY OUTCOMES:
Breast milk composition | up to 6 months
  Influence of diabetes mellitus in the course of pregnancy on the breast milk content of: protein [g/dl], carbohydrates [g/dl], fat [g/dl], energy [kcal/dl].
Adipokines | up to 6 months
  Differences in omentin-1 and visfatin concentrations in serum and breastmilk samples between the study groups.
Impact of maternal adipokines on infantile body fat mass. | up to 6 months
  Correlation of adipokines' concentrations with infantile fat mass will be analysed.
Impact of maternal adipokines on breast milk composition. | up to 6 months
  Correlation of adipokines' concentrations with breast milk content of: protein [g/dl], carbohydrates [g/dl], fat [g/dl], energy [kcal/dl] will be analysed.

CONTACTS AND LOCATIONS:
Locations (1):
- Department and Clinic of Neonatology, Jan Mikulicz-Radecki University Teaching Hospital, Wroclaw Medical University, Wroclaw, Lower Silesian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No